CLINICAL TRIAL: NCT07192575
Title: Enhanced Perioperative Pulmonary Physiotherapy for Prevention of Pulmonary Complications After Laparoscopic Liver Surgery
Brief Title: Prevention of Pulmonary Complications After Laparoscopic Liver Surgery
Acronym: PREPULCION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: Tampere University Hospital (Other); Kuopio University Hospital (Other); University Hospital, Linkoeping (Other); Lund University Hospital (Other)
Responsible Party: Principal Investigator, Minna Nortunen, Md PhD, consultant HPB surgeon, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 254/2023
Record Dates: First submitted 2025-08-25; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Liver Surgery; Pulmonary Complications; Laparoscopic Liver Surgery
Keywords: liver surgery; prehabilitation; pulmonary complications; laparoscopic liver surgery
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: A prospective, multicentre, single-blinded, randomized controlled trial will be conducted according to the study protocol at participating centers. A total of 364 patients scheduled for laparoscopic liver surgery will be randomized at 1:1 ratio into intervention arm or standard ERAS -based perioperative care arm. Block randomization will be used to ensure even distribution of patients with prior pulmonary conditions to both arms. Subgroup analyses will be planned for major/minor liver surgery, pulman
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative pulmonary physiotherapy arm (Active Comparator): Patients in the intervention group receive preoperative breathing education in a single session and an educational video to guide pulmonary training at home. Pulmonary training lasts for 7 days prior to surgery and for 7 days postoperatively. The training includes deep breathing, and coughing, pursed lip breathing and positive expiratory pressure (PEP) therapy. The exercise session (10min) is to be performed two times daily for total of 14 days.
  Interventions: Behavioral: Perioperative Pulmonary Physiotherapy in Laparoscopic Liver Surgery
- Control arm (No Intervention): The control group receives standard perioperative breathing education.

INTERVENTIONS:
Behavioral: Perioperative Pulmonary Physiotherapy in Laparoscopic Liver Surgery — The intervention includes pulmonary physiotherapy training 7 days prior to surgery and 7 days postoperatively. Patients receive physiotherapy education in a single session preoperatively or via an educational video, to guide pulmonary training at home. The pulmonary training includes deep breathing, and coughing, pursed lip breathing and positive expiratory pressure (PEP) therapy. The exercise session (10min) is to be performed two times daily for a total of 14 days.
  Other Names: Pulmonary prehabilitation; Preoprative physiotherapy; Prehabilitation in liver surgery
  Arms: Perioperative pulmonary physiotherapy arm

SUMMARY:
* Background: Postoperative pulmonary complications (PPCs) are the most common complications after major upper abdominal surgery. PPCs include respiratory infections, severe atelectasis, pleural effusion, bronchospasm, aspiration pneumonitis, pneumothorax, exacerbation of chronic pulmonary condition, and respiratory failure. Although PPC rates are higher after open liver surgery, PPCs still occur in approximately 12-13% of patients undergoing laparoscopic liver surgery. Preoperative respiratory physiotherapy education reduces PPCs after open major abdominal surgery and after laparoscopic colorectal surgery. The aim of this study is to investigate the impact of enhanced perioperative pulmonary physiotherapy on the incidence of PPCs after laparoscopic liver surgery.
* Methods: A prospective, multicentre, single-blinded, randomized controlled trial will be conducted according to the study protocol at participating centers. A total of 326 patients scheduled for laparoscopic liver surgery will be randomized at a 1:1 ratio into intervention group or standard Enhanced Recovery After Surgery (ERAS) -based perioperative education group. Surgeons/ researchers are blinded to the patient allocation. Patients in the intervention group receive preoperative breathing education in a single session and an educational video to guide pulmonary training at home. Pulmonary training lasts for 7 days prior to surgery and for 7 days postoperatively. The training includes deep breathing, and coughing, pursed lip breathing and positive expiratory pressure (PEP) therapy. Patients receive instructions for conducting exercises along with an individual risk assessment at a preoperative ambulatory visit. The exercise session (10min) is to be performed two times daily for total of 14 days. The control group receives standard perioperative breathing education. Primary outcome is the rate of postoperative pulmonary complications within 14 days of operation. Secondary outcomes include 90-day mortality, Clavien-Dindo classified complications, length of hospital stay, intensive care unit (ICU) stay, and hospital costs.
* Discussion: Little effort is currently put into preventing pulmonary complications after surgery, although PPCs aggravate considerable morbidity and costs to health care system. ERAS Society protocols concentrate mainly on optimizing postoperative recovery. Laparoscopic techniques as such and frequent manipulation of the diaphragm during liver surgery provoke PPCs at a considerable rate. Aim of the study is to present a short-and-easy perioperative pulmonary physiotherapy initiative and evaluate its impact on PPC rate and PPCs ramifications, including direct costs, after laparoscopic liver surgery.

DETAILED DESCRIPTION:
Background: Postoperative pulmonary complications (PPC) are the most common serious complications after major abdominal surgery. PPC rate varies between 10-50% after open abdominal surgery, depending on the definitions used (Miskovic & Lumb, 2017; PROVE Network Investigators for the Clinical Trial Network of the European Society of Anaesthesiology et al., 2014). According to the European Perioperative Clinical Outcome (EPCO) definition, PPCs enclose clinically relevant pulmonary complications including respiratory infection, atelectasis, pleural effusion, respiratory failure, bronchospasm/ exacerbation of chronic pulmonary condition, pulmonary embolism, aspiration pneumonitis and pneumothorax (Table 1) (Jammer et al., 2015). PPCs cause extensive health care costs due to increased length of stay, ICU days, medication costs, and mortality (Miskovic & Lumb, 2017).

Table 1. Definitions of PPCs (Jammer et al., 2015)

PPCs after abdominal surgery result from shallow breathing due to pain, and abdominal distension, bed rest, long duration of surgery, mucociliary clearance disorder, and dysfunction of diaphragm after mechanical ventilation (Miskovic & Lumb, 2017). Laparoscopic surgery and use of modern Enhanced Recovery After Surgery (ERAS) protocols are associated with reduced PPC rates compared to open surgery, and to poor ERAS compliance (Jurt et al., 2018; Milone et al., 2017). However, PPCs still are the most frequent postoperative complications also after laparoscopic liver surgery, occurring in approximately 12-13% of cases (Fuks et al., 2016; Qin et al., 2021). The relatively high incidence is likely due to laparoscopy and pneumoperitoneum as such, since elevated intra-abdominal pressure accelerates atelectasis formation, decreases respiratory compliance, and causes ventilation/perfusion mismatch, leading to PPCs (Lunardi et al., 2013; Park et al., 2016). PPCs are however more common after laparoscopic liver surgery than after e.g. laparoscopic gastrectomy, where PPC rate is commonly only around 7%(Ntutumu et al., 2016). This implies that specific characteristic of liver surgery, such as manipulation of diaphragm, tendency for postoperative fluid collections under the diaphragm and the disease specific susceptibility of cirrhotic patients for developing PPCs, all most likely affect the higher rate of PPCs after liver surgery.

Different types of interventions have been suggested for preventing PPCs. Preoperative pulmonary physiotherapy education has been shown to reduce PPCs after open major upper abdominal surgery by Boden at al. (Boden et al., 2018). In their RCT of 441 patients, intervention was a single preoperative physiotherapy session, during which the investigators informed the patient about PPCs in general, directed the postoperative physiotherapy exercises, and assessed each patients' individual risk for PPC. The high-quality study showed that this type of small-scale intervention halved the rate of PPCs after open upper abdominal surgery. Cochrane analysis by do Nascimento et al. assessed the effect of incentive spirometry on PPCs compared to no therapy or pulmonary physiotherapy, and found no significant benefit (do Nascimento et al., 2014). Usefulness of perioperative physiotherapy in reducing PPCs after laparoscopic surgery has been studied in two Chinese randomized trials, which both found almost 75% decrease in PPCs in the intervention group (Chen et al., 2022; Qin et al., 2021). The trials were conducted with nearly identical protocols, and by the same research group with patients undergoing laparoscopic colorectal surgery (Qin et al., Chen et al. Clin Rehab 2022). The intervention involved a strenuous, and expensive in-hospital physiotherapy for five days prior to surgery and home-bound pulmonary training for 90 postoperative days.

Prehabilitation programs are recognized as potentially beneficial in avoiding postoperative complications and reducing health care costs (Sliwinski et al., 2023). Protocols in prevention of PPCs are however highly heterogeneous and complex programs and generate a need for extra staff for execution in clinical practice. Research concerning prehabilitation has been criticized for discrepant outcome and methodology measures (Sliwinski et al., 2023), and this also concerns PPC prevention studies. At the moment, no evidence exists on prevention measures to reduce PPCs after any type of laparoscopic upper abdominal surgery. Previous studies on the prevention of PPCs after laparoscopic colorectal surgery present programs that cannot be reasonably integrated to current practices.

Objectives:

The objective of our study is to investigate the effect of a short, perioperative pulmonary physiotherapy (7+7 days) on the incidence of PPCs after laparoscopic liver surgery, in a randomized setting. The control group will receive standard ERAS -protocol based treatment.

Trial design:

The study is a multicenter, randomized controlled trial conducted at five Nordic university hospitals in Finland (Oulu, Tampere, Kuopio) and Sweden (Linköping, Lund). Enrolled subjects will undergo assessments at the following intervals: pre-operative, discharge, and 30 days.

Eligibility criteria:

Inclusion criteria

* Patients who undergo elective, laparoscopic surgery of liver
* Patients able to provide an informed written consent
* Patients capable of completing questionnaires at the time of consent
* Patients compliant in taking in preoperative pulmonary counseling and conducting the exercises

Exclusion criteria

* Age <18 years
* Emergency surgery
* Planned open surgery
* Unwillingness to participate in the follow-up assessment
* No informed consent

Additional consent provisions for collection and use of participant data Data collected within the PREPULCION trial is used only for the purposes determined in the protocol. All modifications to protocol will be communicated with Oulu University Hospital Ethics committee by amendments.

Interventions :

Explanation for the choice of comparators

The main goal in designing the intervention was the direct integrability to current clinical practice, providing the intervention will be shown beneficial. Thus, the intervention followed the crude preoperative path of a patient prepared for major HPB laparoscopy at the Finnish university hospitals. According to current preoperative protocol, patients are scheduled either a visit or a remote appointment at a preoperative outpatient clinic 1-4 weeks prior to surgery. The preoperative clinic visit includes appointments with the surgeon, anesthesiologist, when necessary, preoperative nurse, nutritionist if Nutrition Risk Screening 2002 (NRS2002) score is over 5/13, but no preoperative physiotherapy counseling.

Intervention description

The pulmonary physiotherapy program in the intervention group 7 days pre- and 7 days postoperatively:

I: Thoracic expansion exercises/ diaphragmatic breathing x 10 II: Sustained maximal inspiration, and pursed lip breathing x 10 III: PEP training for 2-3 minutes

IV: Video explaining the pathophysiology of PPCs and instructing all the exercises. preoperatively, at the ward, and after discharge

Hyperlink to the video:

https://api.screen9.com/preview/lSnL3Md0uxXWhO6Xs4A_xVJFomNBwU6TidIydmn_ezjV7iNJtXdRwrpdUyTRu0BO

Criteria for discontinuing or modifying allocated interventions Not applicable.

Strategies to improve adherence to interventions

1. An individual risk assessment (Scholes et al., 2009) can be conducted for each recruited patient during the preoperative outpatient visit if need to improve compliance.
2. A reporting template, where the conducted exercises will be marked pre- and postoperatively, will be provided to patients in the intervention group

   Relevant concomitant care permitted or prohibited during the trial The current perioperative practice at the Finnish university hospitals includes preoperative counseling according to the ERAS recommendations for liver surgery (ERAS Society). ERAS protocols recommend physical prehabilitation, adjusting nutritional status and correcting anemia preoperatively. Pulmonary prehabilitation is not included in the ERAS Societys's recommendations for any gastrointestinal procedures.

   Outcomes

   Primary Outcomes:

   Primary outcome is the incidence of PPCs. PPC is diagnosed according to the study by Scholes et al. (Scholes et al., 2009):

   PPC is diagnosed when four or more of the following criteria were present:
   * Chest radiograph report of collapse/consolidation/ clinically relevant effusion/ edema
   * Raised maximum oral temperature > 38o C on more than one consecutive postoperative day
   * Pulse oximetry oxygen saturation (SpO2) < 90% on more than one consecutive postoperative day
   * Production of yellow or green sputum different to preoperative assessment
   * Presence of infection on sputum culture report
   * An otherwise unexplained white cell count greater than 11 x 109/l or prescription of an antibiotic specific for respiratory infection
   * New abnormal breath sounds on auscultation different to preoperative assessment
   * Physician's diagnosis of postoperative pulmonary complication
   * Presence of pneumonia, bronchitis or clinically relevant effusion/edema on computed chest tomography
   * Presence of pulmonary embolism (PE) on computed chest tomography
   * Exacerbation of chronic pulmonary condition (defined as a need to adjust patient's regular pulmonary medication)

   Secondary outcomes:

   The secondary outcomes are listed below. The mean/median depending on the normality of the outcome will be compared between the groups.
   * Length of stay
   * Use of antibiotics due to a PPC
   * Length of ICU stay
   * Postoperative complications according to Clavien Dindo-classification
   * 90-day mortality
   * Direct hospital costs

   Possible confounders
   * Compliance to perform the planned pulmonary physiotherapy as instructed/ with a correct technique
   * Combining pre- and postoperative interventions
   * Pre-existing pulmonary condition
   * Patient blinding to the intervention is not applicable due to the nature of intervention
   * Investigators will be blinded to ensure non-biased diagnosis of PPCs

   Participant timeline The following data will be recorded prospectively by using specific electronic case report forms (RedCap).

   Baseline
   * Age (at the time of operation)
   * Sex: male - female
   * Charlson Comorbidity Index (CCI): 0, 1, ≥2 (Table 1)
   * NRS2002
   * Body Mass Index (BMI)
   * American Society of Anesthesiologists' Physical Status Classification System (ASA)
   * Clinical Frailty Scale (CFS)
   * anticoagulation if used
   * smoking status/ amount
   * Child-Pugh (digit)
   * pre-existing pulmonary condition, specify
   * Stair-climbing test

   Intervention data
   * type of surgery
   * indication for surgery
   * duration of surgery
   * intraoperative bleeding
   * intraoperative fluid amount/ type
   * intraoperative transfusions
   * mechanical ventilation

     * tidal volume
     * Positive End-Expiratory Pressure (PEEP)
     * Fraction Of Inspired Oxygen (FiO2)
   * use of prophylactic antibiotic
   * use of prophylactic anticoagulation

   Primary hospital stay and discharge
   * PPCs, as diagnosed and defined above
   * All complications during hospital stay measured by Clavien-Dindo classification
   * Re-operations
   * Length of stay (LoS)
   * Discharged to home or another health care unit
   * ICU days
   * Use of antibiotics for PPC

   Sample size According to retrospective patient data from Oulu University Hospital during years 2018-2023, postoperative pneumonia occurred in 11% (23/208) of patients after elective laparoscopic liver resection. The incidence for all PPCs (see the broader definition) is likely higher, but not retraceable retrospectively. In a French retrospective cohort study by Fuks et al, the incidence of all PPCs was 13.2% in the laparoscopic liver resection group. Previous studies with laparoscopic (colorectal) and open upper abdominal procedures have reported a 50-75% reduction in PPCs after enhanced preoperative pulmonary physiotherapy. Accordingly, we estimated the rate of PPCs to 13%, where reduction of 67% would result in 4.3% PPC incidence in the intervention group. When power of 80% and alpha 0.05 are applied, sample size of 326 patients is required. Recruitment is estimated to last from two to three years. We believe that majority of patients are willing to participate, but some drop-outs (estimated as 10%) are expected. Therefore, both groups are designed to include 182 patients with the total sample size of 364 patients.

   All analyses will be performed by or under the guidance of a professional statistician and following the CONSORT guidelines.

   Recruitment All eligible patients will be offered enrolment in the study at the preoperative clinic. A screening log of all elective laparoscopic liver resections throughout the study period is maintained for further assessment of selection biases. After receiving the proper information of the possible advantages and disadvantages of the intervention, and signing the informed consent, the subject will be enrolled. Participating investigators are qualified hepato-pancreatobiliary (HPB) surgeons experienced in the laparoscopic management of liver diseases. Investigators will be blinded for the patient allocation.

   Concealment mechanism Data is collected directly into a digitalized database, REDCap, which is a secure web application for building and managing online databases. It is specifically geared to support online and offline data capture for research studies and operations. Oulu University Hospital ethical committee has approved the level of REDCap data protection.

   Implementation Patients are randomly assigned with a block randomization technique to either an intervention group or control group. Block randomization is performed according to existing pulmonary condition (yes/no) to ensure equal risk of PPCs in both groups. Randomization is performed in a 1:1 ratio according to a computer-generated list compiled by a biostatistician otherwise uninvolved in the clinical care of the trial patients.

   Data collection and management Plans for assessment and collection of outcomes All collected variables are defined in detail in the database. Numbers of missing data will be reported for each variable. The data collection will be the responsibility of the principal investigator and will be reviewed by the study group.

   Data management An electronic database is prospectively maintained throughout the study period. Secure access to the database is granted only to participating investigators. All electronic Case Report Forms (eCRFs) are handled with a special trial idenfication number (ID) and date of birth. Data collected during the study will be stored for 10 years after the publication. Log in history, saved data, and double data entries can be tracked, if necessary. Data ranges are predetermined.

   Confidentiality Patient confidentiality will be strictly maintained. Patients will be assigned a study ID, and all data will be managed without names or personal social security numbers. Access to patient records is limited to the study group and the investigator-delegated study coordinator.

   Plans for collection, laboratory evaluation and storage of biological specimens for genetic or molecular analysis in this trial/future use Not applicable.

   Statistical methods

   Statistical methods for primary and secondary outcomes All analyses will be performed primarily according to the modified intention to treat (ITT) principle, in which all randomized patients are included in the analyses. The primary endpoint will be the incidence of PPCs with 95% confidence interval between the study groups. Secondary outcomes are listed previously. The primary endpoint as well as other categorical data will be analyzed by the χ2-test or Fisher's exact test. Student's t-test or Welch test will be used for continuous variables, the latter if assumption of homogenous variances does not hold.

   Prospectively planned subgroup analyses are listed below. Sample size calculation was performed only for the primary endpoint, and subgroup analyses are hypothesis generating only. The statistical programs SPSS (IBM Corp. Released 2016. IBM SPSS Statistics for Windows, Version 27.0. Armonk, NY: IBM Corp)

   Interim analyses Not required, since no complications can be expected due to the intervention itself.

   Methods for additional analyses (e.g. subgroup analyses) The prospectively planned subgroup analyses are planned and analyzed separately for surgery type (major/minor liver), smoking (yes/no), pre-existing pulmonary condition (yes/no). However, sample size calculation will be done only for the primary endpoint, and subgroup analyses are hypothesis generating only.

ELIGIBILITY:
Inclusion Criteria

* Patients who undergo elective, laparoscopic surgery of liver
* Patients who are able to provide informed written consent
* Patients capable of completing questionnaires at the time of consent
* Patients compliant in taking in preoperative pulmonary counseling and conducting the exercises

Exclusion Criteria:

* Age <18 years
* Emergency surgery
* Planned open surgery
* Unwillingness to participate in the follow up assessment
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative pulmonary complications (PPCs) within 14 days of operation | Complications recorded until 14 days postoperatively
  PPC is diagnosed when four or more of the following criteria were present:
  * Chest radiograph report of collapse/consolidation/ clinically relevant effusion/ edema
  * Raised maximum oral temperature > 38o C on more than one consecutive postoperative day
  * Pulse oximetry oxygen saturation (SpO2) < 90% on more than one consecutive postoperative day
  * Production of yellow or green sputum different to preoperative assessment
  * Presence of infection on sputum culture report
  * An otherwise unexplained white cell count greater than 11 x 109/l or prescription of an antibiotic specific for respiratory infection
  * New abnormal breath sounds on auscultation different to preoperative assessment
  * Physician's diagnosis of postoperative pulmonary complication
  * Presence of pneumonia, bronchitis or clinically relevant effusion/edema on computed chest tomography
  * Presence of pulmonary embolism (PE) on computed chest tomography
  * Exacerbation of chronic pulmonary condition (defined as a need to

SECONDARY OUTCOMES:
Length of stay | 90 days postoperatively
  Length of postoperative hospital stay (days)
Length of intensive care unit (ICU) stay | 90days post operatively
  Length of intensive care unit (ICU) stay (days)
Use of antibiotics postoperatively | 90 days postoperatively
  Use of antibiotics postoperatively, duration, indication, amount and used drug
Postoperative complications | 90 days postoperatively
  Postoperative complications according to Clavien-Dindo
Postoperative mortality | 90days postoperatively
  Postoperative mortality due to any cause
Direct hospital costs | 90 days postoperatively
  Direct hospital cost (euros) of the surgery related stay, including cost of the procedure, length of stay, ICU stay, radiological imaging, reoperations, interventional radiology procedures, laboratory tests and medications.

CONTACTS AND LOCATIONS:
Locations (5):
- Finland (3):
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
- Sweden (2):
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund

IPD SHARING:
Plan to Share IPD: Undecided